CLINICAL TRIAL: NCT00125489
Title: Chloroquine and Sulfadoxine-Pyrimethamine Efficacy for the Treatment of Uncomplicated Falciparum Malaria in Blantyre, Malawi
Brief Title: CQSP in Malawi: Chloroquine and Sulfadoxine-pyrimethamine Efficacy for the Treatment of Malaria in Malawi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0012
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Malaria; Plasmodium Falciparum Malaria
Keywords: chloroquine, malaria, sulfadoxine/pyrimethamine, Malawi
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Chloroquine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: chloroquine sulfate
Drug: sulfadoxine/pyrimethamine

SUMMARY:
The purpose of this research study is to find out how well chloroquine works as a drug to treat malaria in children, compared to the standard malaria treatment in Malawi. In preparation for a longer study of the malaria treatment medication chloroquine alone and in combination with other drugs, a shorter pre-study will be done to compare the anti-malarial effectiveness of chloroquine versus sulfadoxine-pyrimethamine (SP), the standard treatment in Malawi. Two hundred ten children, ages 6 months to 12 years, around Blantyre, Malawi, will be given standard dosing of either chloroquine or SP when they come to the Ndirande Health Centre with signs or symptoms consistent with malaria. The first 30 participants in each treatment group will remain under continuous observation at the health center so that the researchers can monitor their response to the medication until the infection goes away. The participants will be followed for 28 days to see if the the treatment works or fails.

DETAILED DESCRIPTION:
This study follows the observation that chloroquine-resistant malaria may have returned to Malawi, 10 years after its use was eliminated. There is growing consensus that combination chemotherapy should be the rule in malaria treatment to deter the development of drug resistance and possibly also decrease malaria transmission. As sulfadoxine-pyrimethamine (SP) failure rates increase, the reintroduction of chloroquine in Malawi in combination with highly effective rapidly acting drugs such as artesunate and chlorproguanil-dapsone should be considered, and would likely extend the useful life span of each of the drugs. In preparation for a longitudinal clinical trial of chloroquine alone and SP in combination with other drugs, a preliminary trial will be conducted to compare the anti-malarial efficacy of chloroquine versus SP, the standard treatment in Malawi. This is a randomized, open-label clinical trial to compare the antimalarial efficacy of chloroquine versus SP among children with uncomplicated malaria in Blantyre, Malawi. In this study, 210 peri-urban children will be randomly assigned to receive standard dosing of either chloroquine or SP. Follow up will consist of visits on days 2, 3, 7, 14, 21 and 28, according to the standard World Health Organization protocol. Because chloroquine has not been used to treat malaria in Malawi for over a decade, special safety precautions will be taken at the beginning of the study. The first 30 participants in each arm will remain at the Health Centre under continuous observation of the medical staff to monitor response to therapy until they are afebrile for 12 hours and have two consecutive negative 12-hourly blood smears. Observation in an inpatient setting will also help to avoid potential bias due to more intense follow-up of the hospitalized group. A Safety Monitoring Committee (SMC) will meet after the first 30 participants have been enrolled in each arm to determine if the study should stop continuous observation and proceed with out-patient follow up only. All participants will be followed for 28 days to monitor for late therapeutic or parasitologic failure. The primary study objective is to assess the efficacy of chloroquine compared with standard SP therapy, in treating malaria in Malawi, where chloroquine has not been used for over 10 years and to compare it to the efficacy of standard therapy with SP. The secondary study objective is to assess the effect of the re-introduction of chloroquine on the molecular markers associated with chloroquine resistance. The primary study endpoint is the rates of adequate clinical and parasitologic response to therapy. The secondary study endpoints are: (1) rates of early and late therapeutic failure; (2) rates of early and late parasitologic failure; (3) prevalence of chloroquine-resistance conferring pfcrt K76T mutation in pre-treatment infections; (4) rates of pre- and post-treatment pfcrt K76T mutation in cases of chloroquine treatment failure; (5) prevalence of SP-resistance conferring dhfr/dhps mutations in pre-treatment infections; (6) rates of pre- and post-treatment dhfr/dhps mutations in cases of SP treatment failure; (7) clearance time of parasitemia; (8) clearance time of fever; and (9) presence of post-treatment anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >= 6 months to 12 years presenting to Ndirande Health Centre with signs or symptoms consistent with malaria including but not limited to one or more of the following:

   * fever at the time of evaluation (axillary temperature 37.5° C by digital thermometer)
   * report of fever within the last two days
   * profound anemia (conjunctival or palmar pallor)
   * headache
   * body aches
   * abdominal pain
   * decreased intake of food or fluids
   * weakness
2. Positive malaria smear for P. falciparum mono-infection
3. Parasite density of 2,000-200,000/microliter or < 10%
4. Willingness to remain at the Health Centre under continuous observation until the resolution of the infection
5. Parental consent for each participant, and child assent for children older than 5 years

Exclusion Criteria:

1. Signs of severe malaria: One or more of the following:

   * hemoglobin < 5 g/dl
   * parasitemia > 10%
   * prostration * as indicated by inability to drink or breastfeed
   * respiratory distress (deep Kussmaul respirations)
   * bleeding
   * recent seizures*, coma* or mental obtundation* (Blantyre coma score less than 5)
   * persistent vomiting*
2. Presence of a severe disease
3. Presence of a febrile condition caused by diseases other than malaria
4. Known allergy or history of adverse reaction to sulfadoxine/pyrimethamine (SP), sulfa drugs or chloroquine
5. Chronic medication with an antifolate drug
6. Enrollment in this clinical study in the past 28 days *Each of these symptoms or signs is considered a "danger sign."

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210
Dates: Start 2005-05; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Blantyre Malaria Project, Blantyre, Malawi

REFERENCES:
- [Result] Laufer MK, Thesing PC, Eddington ND, Masonga R, Dzinjalamala FK, Takala SL, Taylor TE, Plowe CV. Return of chloroquine antimalarial efficacy in Malawi. N Engl J Med. 2006 Nov 9;355(19):1959-66. doi: 10.1056/NEJMoa062032. PMID 17093247